CLINICAL TRIAL: NCT04952961
Title: Early Detection of Vulval CAncer Through Self-Examination (EDuCATE): Intervention Study A Feasibility Study of Interventions to Promote Vulval Self-examination in Women at Increased Risk of Vulval Cancer
Brief Title: Early Detection of Vulval CAncer Through Self-Examination (EDuCATE): Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: British Society for the Study of Vulval Disease (Unknown)
Responsible Party: Principal Investigator, Vanitha Sivalingam, Academic Clinical Lecturer in Gynaecological Oncology, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 295615
Record Dates: First submitted 2021-06-16; First posted 2021-07-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Self-Examination; Vulvar Cancer; Vulvar Lichen Sclerosus; Vulval Intraepithelial Neoplasia; Vulval Cancer; Vulval Intraepithelial Neoplasia With Lichen Sclerosus; Lichen Planus
MeSH Terms: conditions — Self-Examination; Vulvar Neoplasms; Vulvar Lichen Sclerosus; Lichen Planus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Intervention (Experimental): Participants will be shown how to perform vulval self-examination in a face-to-face intervention and provided with an information leaflet. They will be sent reminders to self-examine each month.
  Interventions: Behavioral: Training in Vulval Self-Examination

INTERVENTIONS:
Behavioral: Training in Vulval Self-Examination — Face-to-face training in vulval self-examination Supplemented with use of aids ( hand mirror, mobile phone with selfie-stick), patient information leaflet, reminders to self-examine

SUMMARY:
Vulval cancer, while rare, has increased in incidence by 17% since the 1990s. It is strongly associated with age, thus this increasing trend is likely to continue with extended life expectancy. Vulval cancer is highly treatable when detected early. Women with chronic vulval conditions including lichen sclerosus, lichen planus and vulval intraepithelial neoplasia are at increased risk of developing vulval cancer. Most patients are in hospital follow-up, however regular vulval self-examination can pick up lesions earlier. There are no formalised methods of teaching self-examination and no evidence that it is acceptable to women.

The main objective of this study is to pilot an intervention to promote and support vulval self-examination for women at increased risk of vulval cancer including those with lichen sclerosus, lichen planus and vulval intraepithelial neoplasia.

Findings from this feasibility study will inform the design of a randomised trial comparing the interventions versus control with an embedded cost-effectiveness analysis.

DETAILED DESCRIPTION:
Vulval cancer is a rare gynaecological cancer, with an increasing incidence rate. IThis trend is expected to risk in years to come because of an aging populating and the increasing rate of human-papillomavirus-related vulval squamous cell carcinoma (VSCC) in young women.

Vulval cancer has a profound effect on the quality of life of women diagnosed with the disease. It carries both disease-related mortality risk and significant morbidity including lower limb lymphoedema, sexual dysfunction and groin discomfort.

Early detection of vulval cancer leads to improved survival and allows for conservative surgical treatment, lower morbidity and improved cosmesis. It is widely agreed that there is no role for screening the general population for vulval cancer; there are no systematic screening programmes nor are there reliable screening methods for identifying malignant precursors . The identification of vulval premalignant and malignant disease, therefore relies on the recognition and reporting of vulval symptoms by the patient and the knowledge and clinical acumen of the health care professional.

There is however, a population of women with chronic vulval conditions who are more likely to develop vulval cancer. Lichen sclerosus (LS), lichen planus (LP) and VIN are recognised precursors of vulval cancer. Regular follow-up in a specialist vulval clinic allows for evaluation of symptom control and treatment compliance and identification of early malignant change; however, regular vulval self-examination may prompt early diagnosis. The interval between noticing a symptom and seeking help could potentially be reduced by providing clear information on signs and symptoms of vulval cancer and guidance on monitoring skin-changes.

Secondary follow-up is not necessary for all women, and women with stable lichen sclerosis are often managed in primary care. Recent guidance from the British Association of Dermatology recommends that women with vulval LS who have responded to treatment be discharged to the care of their general practitioner after a twelve month follow-up period .However, as a majority of women discharged from UK vulval clinics are not subsequently followed up in primary care appropriately, it is important that women are able to self-examine and are confident in recognising and reporting suspicious symptoms. There is, however, no formalised method of teaching vulval self-examination and many women continue with secondary care input.

Self-management focusses on actions that people undertake for themselves to manage their health and illness. In order to self-manage, self-management support is needed (e.g. actions by healthcare professionals). Self-management has been shown to be effective in improving health outcomes such as quality of life. Skin self-examination can reduce mortality in melanoma. A meta-analysis of 18 trials of skin self-examination concluded that interventions including personalised phone counselling, whole body photographs and reminders to perform skin self-examination increased the number of events of patients examining themselves for skin cancer.

A recent mixed-method study by the investigators has demonstrated that only 9% of women have been taught to self-examine, yet up to 86% self-examine regularly. Despite being motivated, 50% reported a lack of confidence in recognition of vulval pathology and a high level of worry about their vulval condition. Both clinicians and patients agreed that face to face teaching was the best intervention for teaching vulval self-examination (unpublished).

The overarching aim of the intervention is to support vulval self-examination in women at high risk of developing vulval cancer. The aims, processes and outcomes were agreed at the focus groups of both women with vulval conditions and clinicians.

The structured intervention will include face-to-face training on vulval self-examination(VSE), supplemented with the use of aids including a hand-mirror or a selfie-stick. Women will be supported with reminders to self-examine, access to a telephone helpline and a leaflet on self-examination.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of a vulval condition with increased risk of malignancy ( lichen sclerosus, lichen planus or vulval intraepithelial neoplasia)
* New diagnosis of a vulval condition with increased risk of malignancy ( lichen sclerosus, lichen planus or vulval intraepithelial neoplasia)
* Must be able to provide informed consent

Exclusion Criteria:

* Inability to consent or complete questionnaires due to cognitive or language issues
* Inability of perform a vulval self-examination due to physical or visual impairments

Note: Those with physical or visual impairments can participate if a dyad is willing to learn how to perform a vulval examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Change in number of self-reported vulval self-examination events | 6 months
  Change in number of self-reported vulval self-examination events over one month before and after the intervention. Patients are asked to record self-examination events in the patient diary

SECONDARY OUTCOMES:
Change in Perceived Vulval Cancer Risk Score | 6 months
  Change in the perceived vulval cancer risk score before and after the intervention. Min 0, Maximum 3. Higher scores indicate higher perceived risk of cancer
Change in Vulval Cancer Worry Scale | 6 months
  This score assesses worry about developing vulval cancer. Change in the score will be assessed before and after the intervention. It has been adapted from the melanoma worry scale. Minimum is 5, Maximum is 19. Higher scores indicate higher worry.
Change in the Hospital anxiety and depression scale | 6 months
  This is a validated scale to measure anxiety and depression in hospital patients. Change will be assessed before and after the intervention. Anxiety and depression can be scored for separately. Minimum score is 0 and Maximum score is 21. Higher scores indicate higher rates of anxiety and depression
Vulval quality of life index | 6 months
  This is a validated measure to assess quality of life in women with vulval disease. Change in the vulval quality of life will be assessed before and after the intervention. Higher scores indicate higher impact of vulval conditions of quality of life. Minimum is 0 and maximum is 45

CONTACTS AND LOCATIONS:
Overall Officials: Vanitha Sivalingam, PhD, Principal Investigator — University of Manchester
Locations (1):
- St Mary's Hospital, Manchester University Hospitals Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No